CLINICAL TRIAL: NCT06124001
Title: An Open-label Phase Ib/IIa Clinical Trial of VG161 Combined With Camrelizumab in the Treatment of Advanced Primary Hepatocellular Carcinoma
Brief Title: Clinical Study of VG161 Combined With Camrelizumab in Patients With Advanced Primary Hepatocellular Carcinoma
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CNBG-Virogin Biotech (Shanghai) Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VG161-C203
Record Dates: First submitted 2023-10-16; First posted 2023-11-09 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Primary Hepatocellular Carcinoma
Keywords: Primary Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — camrelizumab; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Single Arm (Experimental): VG161:
  1)1.0 × 10 ^ 8 PFU daily for 2 consecutive days on Days 1-2 of each cycle (D1-D2); 2)1.0 × 10 ^ 8PFU daily for 3 consecutive days on Days 1-3 of each cycle (D1-D3); camrelizumab: 3 mg/kg every 3 weeks (D8)
  Part2:
  Depends on the recommended dose in Part1
  Interventions: Drug: Recombinant Human IL12/15-PDL1B Oncolytic HSV-1 Injection (Vero Cell)); Drug: camrelizumab for Injection

INTERVENTIONS:
Drug: Recombinant Human IL12/15-PDL1B Oncolytic HSV-1 Injection (Vero Cell)) — Intratumoral injection only. Dosing days may be Days 1-2 or Days 1-3.
  Other Names: VG161
Drug: camrelizumab for Injection — Administered once at 3 mg/kg intravenously on Days 8 of each cycle.
  Other Names: camrelizumab

SUMMARY:
VG161 is a recombinant human-IL12/15/PDL1B oncolytic HSV-1 injection.This study will be conducted in combination with camrelizumab in patients with advanced advanced primary hepatocellular carcinoma who have received at least one first-line treatment regimen. This is an open-label study divided into two parts.

Part 1: This part is an escalating dose trial to explore the safety of the combination and determine the recommended safe dose of the combination.

Part 2: This part is an extension trial to investigate the preliminary efficacy of the combination at a safe dose.

DETAILED DESCRIPTION:
Part1(Phase Ib primary objective): To evaluate the safety and tolerability of VG161 administered by intratumoral injection combined with camrelizumab in the treatment of patients with advanced advanced primary hepatocellular carcinoma who have received at least one first-line treatment regimen. explore the most suitable recommended Phase II dose (RP2D) for combination therapy, and determine the recommended regimen for combination therapy in Phase IIa clinical trials. Secondary objectives:1) Preliminary evaluation of the anti-tumor activity of VG161 combined with camrelizumab in the treatment of patients with advanced primary hepatocellular carcinoma;2) Monitor changes in immunological indicators related to pharmacodynamics;3) Evaluate the impact of herpes simplex virus type I antibody titer levels on the safety and effectiveness of VG161.

Part2(Phase IIa Primary Objective): To evaluate the efficacy of VG161 in combination with carrelizumab in the treatment of patients with advanced primary hepatocellular carcinoma, the main observation index was objective response rate (ORR). Secondary objectives: 1) secondary observations to evaluate the efficacy of combination therapy, including disease control rate (DCR), progression-free survival (PFS), overall survival (OS), and duration of remission (DOR);2) monitoring changes in pharmacodynamic-related immunological indicators;3) To further evaluate the safety of VG161 in combination with carrelizumab.4) To evaluate the effect of herpes simplex virus type I antibody titer level on the safety and efficacy of VG161

ELIGIBILITY:
Inclusion Criteria:

* Subjects must give informed consent to this study before the trial and voluntarily sign a written informed consent form.
* Age 18 to 75 (inclusive), gender is not limited.
* Patients with advanced primary hepatocellular carcinoma confirmed by histopathology or cytology.
* According to the CSCO Guidelines for the Diagnosis and Treatment of Primary Liver Cancer (2022 Edition), patients who have received at least previous first-line treatment regimens that have failed treatment (disease progression or inability to tolerate treatment) must have been treated.
* According to RECIST 1.1, it is determined that at least one CT examination shows that it is measurable and meets the requirements of the volume of injection administration (or the volume of first injection administration in phase IIa) that can be injected under ultrasound guidance (preferably the main tumor burden lesion) under ultrasound guidance, and the longest baseline diameter of the injection lesion (short diameter of lymph node lesions) is >1.5 cm (of which the portal vein lymph node is short, the diameter needs to be > 20 mm).
* Those with positive herpes simplex virus antibody test results (HSV-1 IgG or HSV-1 IgM).
* ECOG physical status score 0-1.
* Estimated survival time of more than 3 months.
* Have adequate organ function:

  1. Routine blood (no blood transfusion or colony-stimulating factor therapy within 14 days): ANC≥ 1.5×109/L, PLT≥75×109/L, Hb≥85g/L, lymphocyte count ≥1.5×109/L (for lymphocyte count 0.8×109/L to 1.5×109/L is determined by the investigator whether to enroll);
  2. Liver function: TBIL≤1.5×ULN, ALT≤5×ULN, AST≤5×ULN;
  3. Child-Pugh A or better B (≤ 7);
  4. Renal function: Cr≤1.5×ULN, and creatinine clearance ≥ 45ml/min (calculated according to Cockcroft-Gault formula);
  5. Coagulation function: activated partial thromboplastin time (APTT) ≤ 1.5×ULN, international normalized ratio (INR) ≤1.5×ULN.
* Eligible subjects of childbearing potential (male and female) must agree to use a reliable method of contraception (hormonal or barrier or abstinence) during the trial and at least 90 days after the last dose (VG161 or carrelizumab, whichever occurs later); Female patients of childbearing age must have a negative blood pregnancy test within 7 days prior to enrollment.

Exclusion Criteria:

* Known fibrolamellar hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma, cholangiocarcinoma or mixed hepatocellular carcinoma.
* Have received chemotherapy, radiotherapy, biological therapy, endocrine therapy, targeted therapy, immunotherapy and other anti-tumor drugs within 4 weeks before the first use of study drugs, among which oral fluorouracils and small molecule targeted drugs are the first use of study drugs. Within the first 2 weeks or the 5 half-lives of the drug (whichever is longer).
* Have received other unmarketed clinical trial treatments within 4 weeks before using the study drug for the first time.
* Have undergone major organ surgery (excluding puncture biopsy) or experienced significant trauma within 4 weeks before taking the study drug for the first time.
* Patients who have received systemic corticosteroids (prednisone >10 mg/day or equivalent doses of similar drugs) or other immunosuppressants within 14 days before the first use of study drugs;Exceptions are the following: treatment with topical, ocular, intraarticular, intranasal, and inhaled corticosteroids; short-term use of corticosteroids (≤10 mg prednisone equivalent) for prophylactic treatment (e.g., prevention of contrast media allergy).
* Have received vaccination within 4 weeks before the first use of study drugs.
* Known severe allergic reaction to any monoclonal antibody.
* The adverse reactions of previous anti-tumor treatments have not returned to CTCAE 5.0 grade ≤1 (except for toxicities such as hair loss that the researcher has judged to have no safety risks).
* Liver tumor burden is greater than 50% of the total liver volume, or those who have received liver transplantation in the past.
* Patients with central nervous system metastasis, spinal cord metastasis and/or spinal cord compression are not suitable for inclusion according to the investigator's judgment.
* In the period of recurrent infection of herpes simplex virus, with corresponding clinical manifestations, such as cold sores, herpetic keratitis, herpetic dermatitis, genital herpes, etc.
* Other uncontrolled active infections.
* Have a history of immunodeficiency, including positive HIV antibody test and positive Treponema pallidum antibody test.
* Patients with active chronic hepatitis B or active hepatitis C (except hepatitis B virus carriers, stable hepatitis B after drug treatment [negative HBV-DNA test or <50IU/ml] and cured hepatitis C patients [HCV RNA Tested negative]).
* Have a history of serious cardiovascular and cerebrovascular diseases:

  1. Ventricular arrhythmias requiring clinical intervention;
  2. QTc interval>480ms;
  3. Acute coronary syndrome, congestive heart failure, stroke or other grade III or above cardiovascular events within 6 months;
  4. New York Heart Association (NYHA) cardiac function class ≥ class II or left ventricular ejection fraction (LVEF) <40%;
  5. Uncontrolled hypertension (systolic blood pressure ≥140mmHg, or diastolic blood pressure ≥90mmHg after treatment).
* Patients with active or past autoimmune diseases that may relapse (such as interstitial pneumonia, colitis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism (including but not limited to these diseases or syndromes, etc.); but does not include patients with clinically stable autoimmune thyroiditis, autoimmune-mediated hypothyroidism treated with a stable dose of thyroid replacement hormone; Type I diabetes on insulin; patients with vitiligo or childhood asthma/allergies that have resolved and do not require any intervention in adulthood.
* Have received immunotherapy and experienced immune-related adverse events (irAEs) such as immune-related pneumonia, myocarditis, etc., which may affect the safety of the trial medication as judged by the researcher.
* Known alcohol or drug dependence.
* People with mental disorders or poor compliance.
* Pregnant or lactating women.
* Patients with obvious symptoms and unstable pleural effusion, peritoneal effusion or pericardial effusion (those with stable clinical symptoms after treatment of pleural effusion, ascites or pericardial effusion can be included).
* The researcher believes that the subject has other serious systemic diseases or other reasons and is not suitable to participate in this clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-11-30 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Phase Ib:RP2D/MTD | through Phase Ib study completion, an average of 8 months
  RP2D/MTD for VG161 in Combination with Camrelizumab
Phase Ib:Incidence and number of DLT | through Phase Ib study completion, an average of 8 months
  Incidence and number of DLT (dose-limiting toxicity)
Phase Ib:AE, SAE occurrence and frequency | through Phase Ib study completion, an average of 8 months
  Occurrence and frequency of AE (Adverse Event) and SAE（Serious adverse event)
Phase IIa:ORR | Time Frame: through Phase IIa study completion, an average of 1 year
  Objective response rate (ORR)

SECONDARY OUTCOMES:
Phase Ib and Phase IIa:ORR | through Phase Ib and Phase IIa study completion, an average of 2 year
  Objective response rate (ORR)
Phase Ib and Phase IIa:DCR | through Phase Ib and Phase IIa study completion, an average of 2 year
  disease control rate (DCR)
Phase Ib and Phase IIa:PFS | through Phase Ib and Phase IIa study completion, an average of 2 year
  Progression Free Survival (PFS)
Phase Ib and Phase IIa:OS | through Phase Ib and Phase IIa study completion, an average of 2 year
  Overall Survival (OS)
Phase Ib and Phase IIa:DOR | through Phase Ib and Phase IIa study completion, an average of 2 year
  Duration of Response (DOR)
Phase Ib and Phase IIa: Immunological indicators | through Phase Ib and Phase IIa study completion, an average of 2 year
  Immunological parameters: peripheral blood lymphocyte subsets (CD3 +, CD4 +, CD8 +, CD4 +/CD8 + ratio, CD19 +,CD16 + CD56 + (NK) cells), cytokines (IL-12, IL-15, IL-6, TNF-α, IFN-γ)
Phase Ib and Phase IIa: herpes simplex virus type I antibodies | through Phase Ib and Phase IIa study completion, an average of 2 year
  Titers of herpes simplex virus type I antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Tingbo Tingbo, MD. PhD., Principal Investigator — Zhejiang University

IPD SHARING:
Plan to Share IPD: No